CLINICAL TRIAL: NCT02528084
Title: The Effects of Yoga on Patients With Rotator Cuff Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Co-Director, Hand and Upper Limb Clinical Research Lab, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB2015
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Rotator Cuff Injuries
Keywords: rotator cuff, shoulder, rehabilitation, yoga
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- yoga intervention (Experimental): patients in the group are asked to follow an online video instructing them various yoga poses. Patients in this group are asked to do the yoga exercises 2-3 times a week, for a total of 6 weeks.
  Interventions: Procedure: yoga
- standard exercises intervention (Experimental): patients in this group are asked to follow an online standard exercises video. Patients in this group are asked to follow specific exercises 2-3 times a day, for a total of 6 weeks.
  Interventions: Procedure: standard exercises
- control (No Intervention): patients in this group carry forth with their daily activities. They are not asked to follow the online yoga video or the online standard exercise video.

INTERVENTIONS:
Procedure: yoga — patients watch and follow an online yoga video.
  Arms: yoga intervention
Procedure: standard exercises — patients watch and follow an online standard exercises video.
  Arms: standard exercises intervention

SUMMARY:
To determine if patients who undergo a 6-week online yoga exercise treatment differ from those who undergo a 6-week online standard exercise intervention and patients who do not undergo any treatment (the control).

DETAILED DESCRIPTION:
Patients awaiting rotator cuff surgery spend months waiting for a doctor's consultation and even longer for surgery. The proposed study is to see if there is a difference between three groups: patients who follow an online yoga video, patients who follow an online standard exercises video and patients who do not undergo either treatment (control).

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old
* rotator cuff injury
* access to YouTube

Exclusion Criteria:

* under 18 years of age
* patient has past yoga experience
* patient will/has undergone any surgery other than rotator cuff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (Pain Level) | 6 weeks
  Shoulder Pain and Disability Index (self-report)
Range of motion (Shoulder Impairment) | 6 weeks
  Shoulder range of motion will be measured using a goniometer (performance-based).

SECONDARY OUTCOMES:
Treatment satisfaction | 6 weeks
  Yes/No question about overall satisfaction (self-report).

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, PhD, Principal Investigator — Western University, Canada; Dolly Mehta, M.Sc., Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided